CLINICAL TRIAL: NCT04993625
Title: Selective Avoidanve of Sentinel Lymph Node Biopsy After Neoadjuvant Chemotherapy In HER-2 Positive/Triple Negative Breast Cancer Patients With Excellent Radiologic Response to the Breast and Axilla, Prospective, Multi-center, Single-arm Study
Brief Title: Selective Avoidance of Sentinel Lymph Node Biopsy After Neoadjuvant Chemotherapy In HER-2 Positive/Triple Negative Breast Cancer Patients With Excellent Radiologic Response to the Breast and Axilla, Prospective, Multi-center, Single-arm (ASLAN) Study
Acronym: ASLAN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jeong Eon Lee (Other)
Collaborators: Seoul National University Hospital (Other); Severance Hospital (Other); Gangnam Severance Hospital (Other); Asan Medical Center (Other)
Responsible Party: Sponsor-Investigator, Jeong Eon Lee, Samsung Medical Center, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2021-02-102
Record Dates: First submitted 2021-07-07; First posted 2021-08-06 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
Keywords: ASLAN
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avoid axillary sentinel lymph node biopsy after neoadjuvant chemotherapy (Experimental)
  Interventions: Procedure: avoid axillary sentinel lymph node biopsy after neoadjuvant chemotherapy

INTERVENTIONS:
Procedure: avoid axillary sentinel lymph node biopsy after neoadjuvant chemotherapy — Selective Omission of Sentinel Lymph Node Biopsy after Neoadjuvant Chemotherapy In HER-2 positive/Triple Negative Breast Cancer Patients with Excellent Radiologic Response to the Breast and Axilla

SUMMARY:
The aims of this study is to evaluate 5 year recurrence free survival when omit sentinel lymph node biopsy after neoadjuvant chemotherapy in triple negative or HER-2 positive breast cancer patients when physical examination expected complete remission. And radiological expected Tumor size ≤ 2cm or non-mass enhancement ≤ 4cm.

ELIGIBILITY:
Inclusion criteria

1. 20≤Age<70
2. undergone neoadjuvant chemotherapy
3. HER-2 or triple negative breast cancer
4. clinical stage T1-3, N0-1, M0 (AJCC 8th)
5. not Inflammatory breast cancer
6. neoadjuvant chemotherapy should be done before surgery(sandwich method is not allowed)

   * least four times anthacycline or taxane-based regimens
   * no axilla lesion progression during chemotherapy
   * no period of adverse response during chemotherapy
7. undergone anti HER-2 therapy in HER-2 positive patient
8. no preoperative anti hormonal therapy
9. no preoperative radiation therapy
10. did not axillary lymph node biopsy before neoadjuvant chemotherapy
11. physical examination expected complete remission. And radiological expected Tumor size ≤ 2cm or non-mass enhancement ≤ 4cm
12. no previous axilla surgery
13. no previous ipsilateral breast surgery for invasive cancer
14. no Pregnancy-associated breast cancer
15. ECOG performance status 0-1
16. Serum or urine b-HCG negative
17. agree to the consent form

Exclusion criteria

1. During pregnancy
2. major depression or taking psychiatric medication
3. significant psychiatric disorder or history of taking antipsychotic drugs
4. any other lymph node metastasis than axillary lesion
5. undergoing total mastectomy
6. do not agree to the consent form

Ages: 20 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
5-year recurrence free survival | 5-year after last patient enrollment
  The aims of this study is to evaluate 5 year recurrence free survival when omit sentinel lymph node biopsy after neoadjuvant chemotherapy in triple negative or HER-2 positive breast cancer patients when expected complete remission.

SECONDARY OUTCOMES:
LRFS | 5-year after last patient enrollment
  5-year local recurrence-free survival
CSS | 5-year after last patient enrollment
  5-year cancer-specific survival
OS | 5-year after last patient enrollment
  5-year overall survival
IBTR | 5-year after last patient enrollment
  5-year ipsilateral breast tumor recurrence interval
IARI | 5-year after last patient enrollment
  5-year ipsilateral axillary recurrence interval
toxicity rate | 5-year after last patient enrollment
  5-year cumulative toxicity rate
EORTC QLQ | 5-year after last patient enrollment
  5-year quality of life
Adverse Event | 5-year after last patient enrollment
  5-year quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Eon Lee, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ryu JM, Lee H, Han W, Lee HB, Ahn SG, Kim HJ, Park HS, Choi JS, Kim H, Cho WK, Lee JE. Selective Avoidance of Sentinel Lymph Node Biopsy After Neoadjuvant Chemotherapy in Human Epidermal Growth Factor 2-Positive/Triple-Negative Breast Cancer Patients With Excellent Response. J Breast Cancer. 2024 Apr;27(2):130-140. doi: 10.4048/jbc.2023.0264. PMID 38685868